CLINICAL TRIAL: NCT06098560
Title: Study on the Clinical Potential of Circulating Tumor DNA in Advanced or Locally Advanced dMMR/MSI-H Colorectal Patients Treated With Immunotherapy
Brief Title: Circulating Tumor DNA (ctDNA) as a Predictive Biomarker for Immunotherapy in Advanced or Locally Advanced dMMR/MSI-H Colorectal Patients
Status: Recruiting | Type: Observational
Sponsor: Geneplus-Beijing Co. Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: PROMISEPLUS-201
Record Dates: First submitted 2023-10-17; First posted 2023-10-24 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Retain tumor tissue samples and series blood samples from each patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
dMMR/MSI-H colorectal cancer patients are the dominant population of immunotherapy/neoadjuvant immunotherapy, but imaging evaluation of immunotherapy efficacy is insufficient. There are some cases, although no disease remission was found on imaging,pathological complete response (pCR) was confirmed after surgery. Meanwhile,previous studies have shown that dynamic changes in ctDNA can help assess immunotherapy efficacy. Therefore, we propose to conduct a multicenter, prospective, observational clinical study to explore the efficacy prediction and monitoring value of ctDNA in immunotherapy for advanced or locally advanced dMMR/MSI-H colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

- advanced or locally advanced dMMR/MSI-H colorectal cancer Expected to receive/be receiving immune checkpoint inhibitor therapy ECOG performance score is 0-1, life expectancy ≥12 weeks

Exclusion Criteria:

- The presence of other uncured malignancies Patients with one or more serious concomitant systemic diseases that, in the investigator's opinion, impair the patient's ability to complete the study Patients with autoimmune disease are not suitable for PD1 monoclonal antibody therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Colorectal cancer patients with MSI-H/dMMR who are expected to receive / receiving immunotherapy
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Correlation of ctDNA changes with pCR rate and the duration of cCR | 2023/12-2025/12
  Correlation of ctDNA changes with rate of pathological complete response or the duration of clinical complete response

SECONDARY OUTCOMES:
Correlation of ctDNA changes with 2 years PFS | 2023/12-2025/12
  Correlation of ctDNA changes with 2 years of progression-free survival after recived immunotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyan Zhou, PhD, Principal Investigator — Fudan University
Locations (2):
- China (2):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Fudan University Shanghai Cancer Center, Shanghai

REFERENCES:
- [Background] Le DT, Durham JN, Smith KN, Wang H, Bartlett BR, Aulakh LK, Lu S, Kemberling H, Wilt C, Luber BS, Wong F, Azad NS, Rucki AA, Laheru D, Donehower R, Zaheer A, Fisher GA, Crocenzi TS, Lee JJ, Greten TF, Duffy AG, Ciombor KK, Eyring AD, Lam BH, Joe A, Kang SP, Holdhoff M, Danilova L, Cope L, Meyer C, Zhou S, Goldberg RM, Armstrong DK, Bever KM, Fader AN, Taube J, Housseau F, Spetzler D, Xiao N, Pardoll DM, Papadopoulos N, Kinzler KW, Eshleman JR, Vogelstein B, Anders RA, Diaz LA Jr. Mismatch repair deficiency predicts response of solid tumors to PD-1 blockade. Science. 2017 Jul 28;357(6349):409-413. doi: 10.1126/science.aan6733. Epub 2017 Jun 8. PMID 28596308
- [Background] Overman MJ, McDermott R, Leach JL, Lonardi S, Lenz HJ, Morse MA, Desai J, Hill A, Axelson M, Moss RA, Goldberg MV, Cao ZA, Ledeine JM, Maglinte GA, Kopetz S, Andre T. Nivolumab in patients with metastatic DNA mismatch repair-deficient or microsatellite instability-high colorectal cancer (CheckMate 142): an open-label, multicentre, phase 2 study. Lancet Oncol. 2017 Sep;18(9):1182-1191. doi: 10.1016/S1470-2045(17)30422-9. Epub 2017 Jul 19. PMID 28734759
- [Background] Overman MJ, Lonardi S, Wong KYM, Lenz HJ, Gelsomino F, Aglietta M, Morse MA, Van Cutsem E, McDermott R, Hill A, Sawyer MB, Hendlisz A, Neyns B, Svrcek M, Moss RA, Ledeine JM, Cao ZA, Kamble S, Kopetz S, Andre T. Durable Clinical Benefit With Nivolumab Plus Ipilimumab in DNA Mismatch Repair-Deficient/Microsatellite Instability-High Metastatic Colorectal Cancer. J Clin Oncol. 2018 Mar 10;36(8):773-779. doi: 10.1200/JCO.2017.76.9901. Epub 2018 Jan 20. PMID 29355075
- [Background] Chalabi M, Fanchi LF, Dijkstra KK, Van den Berg JG, Aalbers AG, Sikorska K, Lopez-Yurda M, Grootscholten C, Beets GL, Snaebjornsson P, Maas M, Mertz M, Veninga V, Bounova G, Broeks A, Beets-Tan RG, de Wijkerslooth TR, van Lent AU, Marsman HA, Nuijten E, Kok NF, Kuiper M, Verbeek WH, Kok M, Van Leerdam ME, Schumacher TN, Voest EE, Haanen JB. Neoadjuvant immunotherapy leads to pathological responses in MMR-proficient and MMR-deficient early-stage colon cancers. Nat Med. 2020 Apr;26(4):566-576. doi: 10.1038/s41591-020-0805-8. Epub 2020 Apr 6. PMID 32251400
- [Background] Dasari A, Morris VK, Allegra CJ, Atreya C, Benson AB 3rd, Boland P, Chung K, Copur MS, Corcoran RB, Deming DA, Dwyer A, Diehn M, Eng C, George TJ, Gollub MJ, Goodwin RA, Hamilton SR, Hechtman JF, Hochster H, Hong TS, Innocenti F, Iqbal A, Jacobs SA, Kennecke HF, Lee JJ, Lieu CH, Lenz HJ, Lindwasser OW, Montagut C, Odisio B, Ou FS, Porter L, Raghav K, Schrag D, Scott AJ, Shi Q, Strickler JH, Venook A, Yaeger R, Yothers G, You YN, Zell JA, Kopetz S. ctDNA applications and integration in colorectal cancer: an NCI Colon and Rectal-Anal Task Forces whitepaper. Nat Rev Clin Oncol. 2020 Dec;17(12):757-770. doi: 10.1038/s41571-020-0392-0. Epub 2020 Jul 6. PMID 32632268